CLINICAL TRIAL: NCT05738187
Title: Evaluation of the Efficacy and Safety of Local Cryotherapy Treatment of Recurrent Head and Neck Cancer in Irradiated Areas: a Pilot Study
Acronym: CRYORL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8761
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Head and Neck Cancer; Local Cryotherapy Treatment
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- local cryotherapy treatment (Experimental)
  Interventions: Procedure: local cryotherapy treatment

INTERVENTIONS:
Procedure: local cryotherapy treatment — cryotherapy

SUMMARY:
In France, squamous cell carcinomas of the head and neck (SCCHN) are the 5th most common cancer. 60% of patients present with locally advanced tumors (stage III/IV), characterized by a poor prognosis (5-year survival not exceeding 60%). The standard treatment consists of either surgical removal followed by adjuvant radiochemotherapy or exclusive radiochemotherapy.

In case of locoregional recurrence (about 40% of patients), salvage surgery can be proposed, allowing prolonged survival for less than one third of eligible patients. However, more than half of locoregional recurrences are unresectable. The standard treatment then consists of immunotherapy and/or chemotherapy for palliative purposes with a median survival of no more than 15 months. Stereotactic radiotherapy is another potentially curative option that allows a local control of 30-60% at 1 year, but at the cost of significant toxicity (up to 50% of grade 3-4 toxicities), thus limiting its indication.

The issue of salvage treatment also applies to other rarer histological forms, including naso-sinus and salivary gland tumors, for which the probability of overall survival at 5 years does not exceed 65% due to locoregional evolution, despite advances in surgical techniques and the addition of radiotherapy.

During the last two decades, minimally invasive interventional radiology techniques have been developed in the field of oncology. Among these techniques, cryotherapy is now commonly used for the treatment of several cancers. The multiplication of its indications is based on numerous clinical advantages (good post-operative analgesia, good toxicity profile, good tumor control). Cryotherapy could thus be a therapeutic alternative in head and neck cancers in recurrence situation in irradiated and unresectable territory, allowing to maintain a curative project in a higher proportion of patients and also to have a more favorable toxicity profile than re-irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Malignant head/neck tumor
* Unresectable locoregional recurrence in a previously irradiated area
* Contraindication to re-irradiation
* Age > 18 years
* Performance index ≤ 2 (WHO)
* Life expectancy > 12 weeks
* Absence of hemostasis disorders
* Renal function: creatinine clearance ≥ 30 mL/min by CKD-EPI method (Cockcroft-Gault formula or MDRD)
* Subject affiliated to a social security health insurance plan
* Subject able to understand the objectives and risks of the research and to give dated and signed informed consent
* For a woman of childbearing age, negative blood pregnancy test at the inclusion visit

Exclusion Criteria:

* Stage IV with distant metastases or multiple tumors
* Melanoma, sarcoma, and lymphoma
* Participants who have received chemotherapy or radiation therapy within 4 weeks
* Other active cancer within the past 2 years (patients with carcinoma in situ, papillary thyroid carcinoma, basal cell skin carcinoma, localized Gleason 6 prostate cancer, or breast cancer in situ are allowed)
* Concomitant therapy with any other systemic anticancer treatment
* Contraindication of anaesthesiology character
* Contraindication to MRI
* Participation in another clinical study
* Any social, medical or psychological condition that may prevent the patient from complying with the constraints of the protocol
* Any significant pathology that may interfere with the patient's participation in the study
* Subject under court protection
* Subject under guardianship or curatorship
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Local tumour control rate | at 12 months
  Tumour control is defined as no increase in size and no suspicious contrast (or radiotracer) in the ablation area. Any suspected recurrence on cross-sectional imaging will be confirmed by biopsy.

SECONDARY OUTCOMES:
Local tumour control rate | at 6 months post-procedure
  Tumour control is defined as no increase in size and no suspicious contrast (or radiotracer) in the ablation area. Any suspected recurrence on cross-sectional imaging will be confirmed by biopsy.
Rate of complications/adverse events (including serious) possibly related to cryotherapy | at 12 months
  assessed by the NCI-CTCAE severity scale version 5.0
To evaluate the quality of life of patients | at 1, 3, 6 and 12 months after cryotherapy
  Scale EORTC-QLQ-C30
To evaluate the quality of life of patients | at 1, 3, 6 and 12 months after cryotherapy
  Scale EORTC - QLQ - H&N35
To evaluate the quality of life of patients | at 1, 3, 6 and 12 months after cryotherapy
  Scale VHI 10
To evaluate the quality of life of patients | at 1, 3, 6 and 12 months after cryotherapy
  Scale MDADI_v1.0
To evaluate the quality of life of patients | at 1, 3, 6 and 12 months after cryotherapy
  Scale DHI

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No